CLINICAL TRIAL: NCT02687789
Title: A Prospective Parallel-design, Double-blind, Randomised, Controlled Investigation to Gain Clinical Experience and Further Knowledge About the Certified Medical Device Vaginal Suppository WO 3191 With Respect to Safety, Tolerability and Efficacy in the Post-Treatment of Bacterial Vaginosis
Brief Title: Safety, Tolerability and Efficacy of Vaginal Suppository WO3191 in the Post-treatment of Bacterial Vaginosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. August Wolff GmbH & Co. KG Arzneimittel (Industry)
Collaborators: PHARMALOG Institute for Clinical Research (Unknown); Bremer Pharmacovigilance Service GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: WOAF-11/2012; CIV-113-12-011731 (Other: EUDRAMED - European Database on Medical Devices)
Record Dates: First submitted 2015-10-12; First posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Vaginosis, Bacterial
Keywords: Bacterial Vaginosis; BV
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical Device: WO3191 (Experimental): The vaginal suppository is used for the reduction and/or inhibition of vaginal biofilms that were shown to be related to recurrent bacterial vaginosis.
  Interventions: Other: Medical Device: WO3191
- Medical Device: Vagisan® Lactic Acid (Active Comparator): It is used for the maintenance and restoration of a natural pH level in the vagina. The acidification of the vaginal milieu with lactic acid promotes the growth of typical vaginal flora (lactic acid bacteria) and is unfavourable for the growth of pathogens in the vagina. Vagisan® Lactic Acid is used in the post-treatment of bacterial vaginosis.
  Interventions: Other: Medical Device: Vagisan® Lactic Acid

INTERVENTIONS:
Other: Medical Device: WO3191 — application of vaginal suppository WO3191: 2 days per week (with a treatment-free interval of three days or two days, respectively; e.g. Monday and Friday)
  Arms: Medical Device: WO3191
Other: Medical Device: Vagisan® Lactic Acid — application of Vagisan® Lactic Acid: 2 days per week (with a treatment-free interval of three days or two days, respectively; e.g. Monday and Friday)
  Arms: Medical Device: Vagisan® Lactic Acid

SUMMARY:
Bacterial Vaginosis (BV) is a common infectious disorder and is characterized by a disturbance in the vaginal microbiological milieu. Anaerobic bacteria, such as Gardnerella vaginalis and Atopobium vaginae overgrow the physiologic vaginal flora which is dominated by Lactobacilli. BV can arise and remit spontaneously but often presents as a recurrent disease.

New findings indicate that the presence of an adherent bacterial biofilm on the vaginal mucosa seems to be the reason for the recurrence of BV as well as the overgrowth condition by anaerobic bacteria. Biofilms are defined as a structured consortium of bacteria embedded in a matrix of extracellular polymeric substances (EPS).

The purpose of this study is to achieve substantial results with respect to tolerability and safety, and to gain further knowledge on the clinical efficacy of Vaginal suppository WO3191, the investigation will be performed in a parallel-design, double-blind, randomised, controlled manner.

DETAILED DESCRIPTION:
This investigation is a multicentre, parallel-group, double-blind, controlled trial with an open Follow-up Phase of 12 weeks. It is conducted to gain clinical experience and further knowledge about the certified medical device Vaginal suppository WO3191 in women with bacterial vaginosis.

In this investigation the Investigational Medical Device (IMD) will be used as post-treatment following standard therapy with oral metronidazole for BV. IMD will be applied 2 times a week for 3 weeks.

The primary purpose is the evaluation of the safety and local tolerability of WO3191, therefore all adverse events (AEs) and adverse device effects (ADEs) will be documented. Furthermore, patients will be asked for possibly arising subjective vaginal symptoms (burning, itching, bleeding, pain, dryness) and will be examined for possibly arising objective vaginal findings (redness, petechial bleeding, dryness, swelling).

The secondary purpose of this investigation is to gain clinical experience and further knowledge about Vaginal suppository WO3191 with respect to the efficacy in the post-treatment of bacterial vaginosis.

In addition pH-values and microbiological data shall be examined.

Furthermore, the difference between Vaginal suppository WO3191 (Group A) and the comparator (Vagisan® Lactic Acid, group B) with respect to the safety, tolerability and the efficacy in the post-treatment of bacterial vaginosis shall be evaluated exploratively.

Patients who have completed all regular visits (Visit 1 - 4; Visit 1 - Screening, Visit 2 - Randomization, Start of application of IMD; Visit 3 - one week after Visit 2; Visit 4 - two weeks after Visit 3, End of application of IMD) of the investigation shall attend an observational Follow-up Phase of 12 weeks with a final Visit 5. At Visit 5 recurrences of BV as well as the sustainability of the efficacy of Vaginal suppository WO3191 will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Signed declaration of consent and signed data protection declaration after having been informed about the nature, relevance and the scope of the investigation and about the expected desired and undesired effects of the IMD
* Premenopause, age 18 to 50 years (incl. patients with Intrauterine device, e.g. Mirena® with amenorrhoea)
* Acute BV (at least 3 of 4 Amsel's Criteria fulfilled and Nugent Score > 6)
* Existing bacterial biofilm in the vagina, verified by positive EPS of bacterial biofilm and by microscopy
* Requirement of oral treatment of metronidazole for BV

Exclusion Criteria:

* Postmenopause (no menses in the last six months prior to enrolment)
* Positive Herpes simplex infection
* Positive Candida spp. infection
* Positive Trichomonas spp. infection
* Pathologic PAP (III, III D-V) within the last 3 months
* Chronic immunosuppressive diseases (i.e. HIV) or treatment (i.e. transplantation)
* Malignant conditions of CIN, VIN or VAIN, currently and / or within the past 6 months
* Presence or history (within the last 5 years) of any other malignancy
* Previous chemotherapy (within 6 months before start of this investigation)
* Current vaginal or systemic treatment with antibiotics or corticosteroids, systemic treatment with NSAIDs (nonsteroidal anti-inflammatory drugs) within the last two weeks prior to start of this investigation (except metronidazole for the treatment of BV: prescription of metronidazole before investigation entry; except NSAIDs taken in a single dose in case of need, e.g. for headache)
* Use of not permitted contraception or not willing to use contraception (Allowed contraception: oral hormonal contraceptives, intrauterine device, surgical, sexual abstinence; Not permitted contraception: condoms, local spermicides, intravaginal contraceptive measures)
* Pregnancy or lactation
* Active Smokers (more than 5 cigarettes per day)
* Use of any other intravaginal medicinal product or medical device (including all intravaginal contraceptive measures (e.g. NuvaRing®, local spermicides)
* Known hypersensitivity to one or more of the active and / or inactive ingredients of the antibiotic treatment (metronidazole: mandatory for inclusion)
* Known hypersensitivity to one or more of the ingredients of the IMD (test product and/or comparator)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Local tolerability of IMD defined as a cumulative sum score of solicited local ADE for each Patient | 3 weeks
  Local tolerability of the IMD will be defined as a cumulative sum score of the solicited local (vaginal) ADE (consisting of subjectively experienced symptoms rated by the patient: burning, itching, bleeding, pain, dryness and objectively documented findings rated by the physician: redness, petechial bleeding, dryness, swelling) for each patient after 1 and 3 weeks of application (Visit 3 and Visit 4, respectively).

SECONDARY OUTCOMES:
Subjective symptoms (local tolerability) | 3 weeks
  Each of the subjective symptoms (scored from 0 [none/normal] to 3 [severe]) at Visit 2 (before the first application), Visit 3 (after 1 week of application) and Visit 4 (after 3 weeks of application)
Objective findings | 3 weeks
  Each finding (scored from 0 [none/normal] to 3 [severe]) as well as each sum score at Visit 3 (after 1 week of application) and Visit 4 (after 3 weeks of application) will be summarised by the maximum value and the mean value for Visit 3 and Visit 4, respectively
Global judgement of tolerability | 3 weeks
  Global judgement of tolerability by investigator and patient at Visit 4 (after 3 weeks of application)
AE and ADE (Safety) | up to 4 months
  Unsolicited AEs and ADEs
Occurrence of AE / SAE / ADE / SADE (Serious Adverse Event) (Safety) | up to 4 months
  Occurrence of AE / SAE / ADE / SADE
Characteristics of AE / SAE / ADE / SADE (Safety) | up to 4 months
  Characteristics of occured AE / SAE / ADE / SADE
Change in biofilm EPS | up to 4 months
  Proof of the biofilm EPS at Visit 2 (before the first application), Visit 3 (after 1 week of application), Visit 4 (after 3 weeks of application) and Visit 5 (after Follow-up Phase, i.e.12 weeks after the end of the application Phase (Visit 4))
  Combined Parameter: Evaluation of Extracellular Polymeric Substances (EPS) in urine samples and evaluation of existence of bacterial biofilm
Change in pH-value from vaginal smear | within 4 months
  pH-value from vaginal smear at visit 2 (before the first application), Visit 3 (after 1 week of application), Visit 4 (after 3 weeks of application) and Visit 5 (after Follow-up Phase, i.e.12 weeks after the end of the application Phase (Visit 4))
Change in Nugent-Score | within 3 weeks
  Nugent-Score at Visit 2 (before the first application), Visit 3 (after 1 week of application) and Visit 4 (after 3 weeks of application)
Change in Vaginal flora | within 4 months
  Vaginal flora (Lactobacillus spp., Atopobium vaginae and Gardnerella vaginalis) at Visit 2 (before the first application), Visit 3 (after 1 week of application) Visit 4 (after 3 weeks of application) and Visit 5 (after Follow-up Phase, i.e.12 weeks after the end of the application Phase (Visit 4))
Time to recurrence of BV | up to 3 months
  Time from the end of application (Visit 4) to the first recurrence of BV within the Follow-up Phase of 12 weeks

OTHER OUTCOMES:
Global judgement of the IMD | 3 weeks
  Global judgement of the IMD by investigator and patient

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Christoph Abels, MD, Study Director — Dr. August Wolff GmbH & Co. KG Arzneimittel; Prof. Werner Mendling, MD, Principal Investigator — St. Anna Klinik, Wuppertal
Locations (13):
- Germany (13):
  - Dr. Gerick, Aachen
  - Dr. Hofmann, Betzdorf
  - Dr. de Brabandt, Bielefeld
  - Dr. Werner Göttker-Schnetmann, Frankfurt
  - Dr. Deininger, Munich
  - Dr. Kränzlin, Munich
  - Dr. Kästner, Munich
  - Dr. Kühne, Munich
  - Bianca Moll-Bosch, Siegen
  - Dr. Susanne Feidicker, Steinhagen
  - Thomas Riepen, Weilburg
  - Dr. Waldschütz, Wuppertal
  - Prof. Mendling, Wuppertal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gottschick C, Deng ZL, Vital M, Masur C, Abels C, Pieper DH, Rohde M, Mendling W, Wagner-Dobler I. Treatment of biofilms in bacterial vaginosis by an amphoteric tenside pessary-clinical study and microbiota analysis. Microbiome. 2017 Sep 13;5(1):119. doi: 10.1186/s40168-017-0326-y. PMID 28903767
- [Derived] Gottschick C, Deng ZL, Vital M, Masur C, Abels C, Pieper DH, Wagner-Dobler I. The urinary microbiota of men and women and its changes in women during bacterial vaginosis and antibiotic treatment. Microbiome. 2017 Aug 14;5(1):99. doi: 10.1186/s40168-017-0305-3. PMID 28807017